CLINICAL TRIAL: NCT01238159
Title: Open-labeled, Multicenter Phase II Study of Concomitant Chemo-radiotherapy Followed by MIDLE (Methotrexate, Ifosfamide, Dexamethasone, L-asparaginase, Etoposide) Chemotherapy in Stage I/II Extranodal NK/T-cell Lymphoma
Brief Title: Concomitant Chemo-radiotherapy Followed by MIDLE Chemotherapy in Stage I/II Extranodal NK/T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Asan Medical Center (Other); Yonsei University (Other); Seoul National University (Other); Chonnam National University (Other)
Responsible Party: Principal Investigator, Kim, Seok Jin, Associate professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-06-019
Record Dates: First submitted 2010-09-08; First posted 2010-11-10 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Extranodal NK-T-Cell Lymphoma, Nasal and Nasal-Type
Keywords: Natural killer cell; T cell; Lymphoma; Radiation; Chemotherapy
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CCRT+MIDLE (Experimental): Patients who are planned to be treated with CCRT plus MIDLE chemotherapy. CCRT means concurrent chemoradiation, and MIDLE represent systemic chemotherapy.
  Interventions: Radiation: CCRT+MIDLE chemotherapy

INTERVENTIONS:
Radiation: CCRT+MIDLE chemotherapy — Patients are planned to be treated with CCRT plus MIDLE chemotherapy
  Other Names: Chemoradiotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy of concomitant chemoradiation followed by MIDLE chemotherapy for stage I/II extranodal NK/T cell lymphoma.

DETAILED DESCRIPTION:
Concomitant chemo-radiotherapy:

Radiation 36-44 Gy/18-22 fractions (2 Gy/fraction) Weekly Cisplatin 30mg/m2 + N/S 100ml MIV over 30min Tri-weekly L-asparaginase 4000 IU IV (D1, 3, 5)

Rest period: 3 weeks

MIDLE chemotherapy: Repeated every 28 days for 2 cycles D1 Methotrexate 3g/m2 + D5W 500ml MIV over 6 hours D2-D3 Etoposide 100mg/m2 + D5W 500ml MIV over 90mins D2-D3 Ifosfamide 1000mg/m2 + D5W 100ml MIV over 1hr D2-D3 Mesna 300mg/m2 + D5W 100ml MIV over 15mins (-15min, 4hrs and 8hrs after ifosfamide, total 3 doses) D1-D4 Dexamethasone 40mg/d PO or IV D4, 6, 8, 14, 10 L-asparaginase 6000IU/m2 + D5W 500ml MIV over 2hours

ELIGIBILITY:
Inclusion Criteria:

* patients were required to have a biopsy-proven diagnosis of nasal ENKTL
* at least 18 years old
* Ann Arbor stage IE or IIE
* measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 life expectancy greater than 12 weeks
* adequate hematologic (hemoglobin > 9.0 g/dL, absolute neutrophil count > 1,500/uL and platelets > 100,000/uL)
* renal (serum creatinine < 1.5 mg/dL, creatinine clearance > 50 mL/min)
* hepatic (total bilirubin < 2 times of upper limit of normal and aspartate transferase < 3 times of upper limit of normal) function
* Diagnosis of ENKTL is based on the presence of histological features and immunophenotypes compatible with ENKTL (e.g., cytoplasmic CD3+, CD20-, CD56+,
* positive for cytotoxic molecules
* positive for EBV by in situ hybridization).
* Informed consent

Exclusion Criteria:

* prior or concomitant malignant tumors
* any coexisting medical problems of sufficient severity to prevent full compliance with the study protocol.
* ENKTL with non-nasal sites such as skin or gastrointestinal tract was excluded even if it is localized.
* Other subtypes of non-Hodgkin lymphoma (NHL), including myeloid/NK cell precursor acute leukemia, blastic NK cell lymphoma/precursor NK cell lymphoblastic leukemia, aggressive NK cell leukemia, and peripheral T cell lymphoma, unspecified, were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Complete response | Within 4 weeks after the completion of planned treatment
  The response criteria was based on the International Working Group Report (1999).

SECONDARY OUTCOMES:
Overall response rate | Up to 2 years
  Overall response rate includes complete and partial response.
overall survival | up to 2 years
  Overall survival is defined as the time interval between the date of diagnosis and the date of death with any cause.
Progression-free survival | up to 2 years
  Progression-free survival is defined as the time interval between the the date of diagnosis and the date of death with any cause or disease progression/relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea